CLINICAL TRIAL: NCT04048135
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetic Properties of BIO89-100 Administered Subcutaneously in Subjects With Nonalcoholic Steatohepatitis (NASH) or With Nonalcoholic Fatty Liver Disease (NAFLD) and at High Risk of NASH
Brief Title: A Multiple Ascending Dose Study of Pegozafermin in Participants With Biopsy Confirmed Nonalcoholic Steatohepatitis (NASH) or Nonalcoholic Fatty Liver Disease (NAFLD) and at High Risk of NASH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Collaborators: ProSciento, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO89-100-002
Record Dates: First submitted 2019-08-04; First posted 2019-08-07 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-02

CONDITIONS: NASH
Keywords: NASH, NAFLD; Liver diseases; Fatty Liver; Metabolic diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 was blinded, Part 2 was open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Pegozafermin 3 milligrams (mg) weekly (QW) (Experimental): Participants were administered 3 mg of pegozafermin QW, via subcutaneous (SC) injection, starting on Day 1 through Day 85.
  Interventions: Drug: Pegozafermin
- Part 1: Pegozafermin 9 mg QW (Experimental): Participants were administered 9 mg of pegozafermin QW, via SC injection, starting on Day 1 through Day 85.
  Interventions: Drug: Pegozafermin
- Part 1: Pegozafermin 18 mg QW (Experimental): Participants were administered 18 mg of pegozafermin QW, via SC injection, starting on Day 1 through Day 85.
  Interventions: Drug: Pegozafermin
- Part 1: Pegozafermin 27 mg QW (Experimental): Participants were administered 27 mg of pegozafermin QW, via SC injection, starting on Day 1 through Day 85.
  Interventions: Drug: Pegozafermin
- Part 1: Pegozafermin 18 mg Every 2 Weeks (Q2W) (Experimental): Participants were administered 18 mg of pegozafermin Q2W, via SC injection, starting on Day 1 through Day 85.
  Interventions: Drug: Pegozafermin
- Part 1: Pegozafermin 36 mg Q2W (Experimental): Participants were administered 36 mg of pegozafermin Q2W, via SC injection, starting on Day 1 through Day 85.
  Interventions: Drug: Pegozafermin
- Part 1: Placebo QW or Q2W (Placebo Comparator): Participants were administered placebo matching to pegozafermin QW or Q2W, via SC injection, starting on Day 1 through Day 85.
  Interventions: Other: Placebo
- Part 2: Pegozafermin 27 mg QW (Experimental): Participants were administered 27 mg of pegozafermin QW, via SC injection, starting on Day 1 through Day 134.
  Interventions: Drug: Pegozafermin

INTERVENTIONS:
Drug: Pegozafermin — Subcutaneous injection
  Other Names: BIO89-100
  Arms: Part 1: Pegozafermin 18 mg Every 2 Weeks (Q2W); Part 1: Pegozafermin 18 mg QW; Part 1: Pegozafermin 27 mg QW; Part 1: Pegozafermin 3 milligrams (mg) weekly (QW); Part 1: Pegozafermin 36 mg Q2W; Part 1: Pegozafermin 9 mg QW; Part 2: Pegozafermin 27 mg QW
Other: Placebo — Subcutaneous injection
  Arms: Part 1: Placebo QW or Q2W

SUMMARY:
Part 1: This is a multi-center evaluation of pegozafermin (administered weekly or every other week) in a randomized, double-blind, placebo-controlled study administered for 12 weeks in participants with NASH and NAFLD at high risk of NASH, including a pre-defined number of participants with biopsy confirmed NASH and fibrosis stages F1-F3 to be enrolled.

Part 2: This is a multi-center, open label evaluation of pegozafermin at 27 mg administered weekly for 20 weeks in participants with biopsy-proven NASH (NAS ≥4, fibrosis stage F2 or F3).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be 21 to 75 years of age inclusive, at the time of signing the informed consent form (ICF).
* Evidence of steatosis by Fibroscan and magnetic resonance imaging based proton density fat fraction (MRI-PDFF)
* NASH or NAFLD at high risk for NASH as reflected by AT LEAST ONE of the following:
* Diagnosis of NASH with fibrosis (stages F1, F2 or F3), without cirrhosis, by percutaneous liver biopsy within 24 months prior to screening
* Central obesity WITH type 2 diabetes mellitus (T2DM)
* Central obesity WITH either increased alanine transaminase (ALT) and/or Fibroscan vibration-controlled transient elastography (VCTE) score ≥7 KPa.
* Part 2 only: Biopsy-proven NASH in a liver biopsy obtained within 24 weeks of baseline with fibrosis stage F2 or F3 and NAS ≥4, with a score of at least 1 in each of steatosis, ballooning degeneration, and lobular inflammation. A small number of high risk F1 allowed.

Key Exclusion Criteria:

* Clinically significant disorder or a history of any illness that, in the opinion of the Investigator, might confound the results of the study, or pose additional risk to the participant by participation in the study.
* History of type 1 diabetes.
* Weight loss of more than 5% within 3 months prior to Day -1 or more than 10% within 6 months prior to Day -1 or planning to try to lose weight during conduct of study.
* History of a liver disorder other than NASH or clinical suspicion of a liver disorder other than NASH
* History of cirrhosis or evidence of cirrhosis

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlton, MD, Study Director — 89bio, Inc.
Locations (25):
- United States (24):
  - 89bio Clinical Study Site, Madison, Alabama
  - 89bio Clinical Study Site, Chandler, Arizona
  - 89bio Clinical Study Site, Tucson, Arizona
  - 89bio Clinical Study Site, Chula Vista, California
  - 89bio Clinical Study Site, Huntington Beach, California
  - 89bio Clinical Study Site, Montclair, California
  - 89bio Clinical Study Site, Miami, Florida
  - 89bio Clinical Study Site, Miami Lakes, Florida
  - 89bio Clinical Study Site, Ocala, Florida
  - 89bio Clinical Study Site, Sarasota, Florida
  - 89bio Clinical Study Site, Lake Charles, Louisiana
  - 89bio Clinical Study Site, Berlin, New Jersey
  - 89bio Clinical Study Site, Florham Park, New Jersey
  - 89bio Clinical Study Site, East Syracuse, New York
  - 89bio Clinical Study Site, Concord, North Carolina
  - 89bio Clinical Study Site, Raleigh, North Carolina
  - 89bio Clinical Study Site, Greenwood, South Carolina
  - 89bio Clinical Study Site, Summerville, South Carolina
  - 89bio Clinical Study Site, Hermitage, Tennessee
  - 89bio Clinical Study Site, Austin, Texas
  - 89bio Clinical Study Site, Edinburg, Texas
  - 89bio Clinical Study Site, Houston, Texas
  - 89bio Clinical Study Site, San Antonio, Texas
  - 89bio Clinical Study Site, Wichita Falls, Texas
- 89bio Clinical Study Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alkhouri N, Lazas D, Loomba R, Frias JP, Feng S, Tseng L, Balic K, Agollah GD, Kwan T, Iyer JS, Morrow L, Mansbach H, Margalit M, Harrison SA. Clinical trial: Effects of pegozafermin on the liver and on metabolic comorbidities in subjects with biopsy-confirmed nonalcoholic steatohepatitis. Aliment Pharmacol Ther. 2023 Nov;58(10):1005-1015. doi: 10.1111/apt.17709. Epub 2023 Sep 18. PMID 37718721
- [Derived] Tseng CL, Balic K, Charlton RW, Margalit M, Mansbach H, Savic RM. Population Pharmacokinetics and Pharmacodynamics of Pegozafermin in Patients with Nonalcoholic Steatohepatitis. Clin Pharmacol Ther. 2023 Dec;114(6):1323-1331. doi: 10.1002/cpt.3046. Epub 2023 Oct 2. PMID 37696614
- [Derived] Loomba R, Lawitz EJ, Frias JP, Ortiz-Lasanta G, Johansson L, Franey BB, Morrow L, Rosenstock M, Hartsfield CL, Chen CY, Tseng L, Charlton RW, Mansbach H, Margalit M. Safety, pharmacokinetics, and pharmacodynamics of pegozafermin in patients with non-alcoholic steatohepatitis: a randomised, double-blind, placebo-controlled, phase 1b/2a multiple-ascending-dose study. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):120-132. doi: 10.1016/S2468-1253(22)00347-8. Epub 2022 Dec 12. PMID 36521501
- See also: Related Info — https://doi.org/10.1016/S2468-1253(22)00347-8

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1: Pegozafermin 3 Milligrams (mg) Weekly (QW) | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Every 2 Weeks (Q2W) | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W | Part 2: Pegozafermin 27 mg QW
Started | 6 | 12 | 11 | 10 | 14 | 9 | 19 | 20
Received 1 Dose of Study Drug (Randomized Analysis Set. Arm groups were based upon planned treatment.) | 6 | 12 | 11 | 10 | 14 | 9 | 19 | 20
Safety Analysis Set (Arm groups were based upon the actual treatment received for the purpose of safety analysis.) | 7 (One participant was randomized to the placebo group but received a single dose of pegozafermin 3 mg instead.) | 12 | 11 | 10 | 14 | 9 | 18 (One participant was randomized to the placebo group but received a single dose of pegozafermin 3 mg instead.) | 20
Completed | 5 | 11 | 10 | 7 | 13 | 8 | 18 | 19
Not Completed | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population description: For Part 1, randomized analysis set included all randomized participants who received at least 1 dose of investigational product. For Part 2, Full analysis set included all enrolled participants who received at least 1 dose of investigational product.
Groups:
- Part 1: Pegozafermin 3 mg QW: Participants were administered 3 mg of pegozafermin QW, via SC injection, starting on Day 1 through Day 85.
- Part 1: Pegozafermin 18 mg Q2W: Participants were administered 18 mg of pegozafermin Q2W, via SC injection, starting on Day 1 through Day 85.
- Total: Total of all reporting groups
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W | Part 2: Pegozafermin 27 mg QW | Total
Number analyzed (Participants) | 6 | 12 | 11 | 10 | 14 | 9 | 19 | 20 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.13 (8.23) | 49.50 (11.45) | 51.47 (13.39) | 51.96 (9.83) | 51.22 (8.14) | 52.46 (8.73) | 52.62 (8.99) | 58.44 (9.07) | 52.97 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 8 | 10 | 1 | 12 | 15 | 65
  Male | 1 | 6 | 3 | 2 | 4 | 8 | 7 | 5 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 9 | 10 | 13 | 9 | 16 | 5 | 79
  Not Hispanic or Latino | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 15 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 5
  White | 5 | 11 | 9 | 10 | 13 | 9 | 17 | 20 | 94
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-emergent Adverse Event (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were defined as AEs occurring at or after the first dose date and time, through study termination, or existing prior to the time of and worsening after the time of the first dose of investigational product. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to 113 days
Population: The Safety Analysis set included all randomized participants who received at least 1 dose of study intervention. Arm groups were based upon the actual treatment received for the purpose of safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W
Number analyzed (Participants) | 7 | 12 | 11 | 10 | 14 | 9 | 18
Participants | 6 | 4 | 7 | 7 | 8 | 8 | 8

2. Primary Outcome: Part 2: Number of Participants With TEAEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were defined as AEs occurring at or after the first dose date and time, through study termination, or existing prior to the time of and worsening after the time of the first dose of investigational product. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to 162 days
Population: The Full Analysis Set included all enrolled participants in Part 2 who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 20
Participants | 18

3. Primary Outcome: Part 1: Maximum Observed Serum Concentration (Cmax) of Pegozafermin
Time Frame: Predose and up to 168 hours postdose on Day 29
Population: The PK Analysis set included all randomized participants who received at least 1 dose of study intervention and had at least 1 on-study PK measurement.
Measure: Median (90% Confidence Interval); unit: ng/mL
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W
Number analyzed (Participants) | 6 | 12 | 11 | 10 | 14 | 9
ng/mL | 103 [59 to 156] | 439 [238 to 852] | 901 [200 to 1281] | 1166 [566 to 2243] | 649 [160 to 1300] | 1674 [1300 to 2791]

4. Primary Outcome: Part 1: Area Under the Serum Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUClast) of Pegozafermin
Time Frame: Predose and up to 168 hours postdose on Day 29
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: ng*hour/mL
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W
Number analyzed (Participants) | 6 | 12 | 11 | 10 | 14 | 9
ng*hour/mL | 11879 [7350 to 17778] | 42576 [24394 to 70300] | 95765 [24822 to 138904] | 112632 [57880 to 231937] | 78761 [20520 to 155994] | 209436 [153404 to 287414]

5. Primary Outcome: Part 1: Time to Peak Serum Concentration (Tmax) of Pegozafermin
Time Frame: Predose and up to 168 hours postdose on Day 29
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: hr
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W
Number analyzed (Participants) | 6 | 12 | 11 | 10 | 14 | 9
hr | 59.5 [47.3 to 72.0] | 48.0 [18.6 to 58.8] | 48.0 [34.7 to 72.1] | 48.1 [46.3 to 63.4] | 72.0 [47.5 to 95.2] | 48.0 [45.2 to 71.6]

6. Primary Outcome: Part 1: Terminal Elimination Half-life (t1/2) of Pegozafermin
Time Frame: Predose and up to 168 hours postdose on Day 29
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: hr
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W
Number analyzed (Participants) | 6 | 12 | 11 | 10 | 14 | 9
hr | 57.1 [54.0 to 75.3] | 46.3 [36.1 to 67.7] | 68.1 [50.8 to 114.0] | 53.0 [27.9 to 62.2] | 54.4 [45.5 to 70.4] | 53.2 [37.4 to 62.2]

7. Primary Outcome: Part 2: Number of Participants With at Least a 2-point Improvement in NAFLD Activity Score (NAS) With at Least a 1-point Improvement in Ballooning or Lobular Inflammation, and no Worsening of Fibrosis
Description: NAS was the sum of the scores of steatosis, inflammation, and ballooning. NAS score ranges from of 0 to 8, with higher scores indicating worse disease severity.
  Worsening of fibrosis was defined as progression of fibrosis ≥1 stage in NASH Clinical Research Network (CRN) fibrosis score.
  NASH CRN Fibrosis is staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: Day 141
Population: The Histology Biopsy Analysis Set included all enrolled participants who received at least 1 dose of study intervention and who had both baseline (screening or eligible historical) and post-baseline biopsies.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 19
Participants | 12

8. Secondary Outcome: Part 1: Number of Participants With a Positive Anti-Drug Antibodies (ADA) Response to Pegozafermin
Description: Number of participants with anti-pegozafermin antibodies (ADA) with status as ADA positive has been reported.
Time Frame: Up to 113 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W
Number analyzed (Participants) | 7 | 12 | 11 | 10 | 14 | 9 | 18
Participants | 1 | 9 | 7 | 7 | 11 | 6 | 2

9. Secondary Outcome: Parts 1 and 2: Percent Change From Baseline in Body Weight
Description: Least Squares (LS) Mean was calculated using mixed-model repeated measures (MMRM).
Time Frame: Part 1: Baseline, Day 85; Part 2: Baseline, Day 141
Population: The analysis set included all randomized participants who received at least 1 dose of study intervention and who had measurable post-baseline PD data in Parts 1 and 2. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 5 | 11 | 10 | 7 | 13 | 8 | 18 | 19
Percent change | 1.19 (1.06) | 2.59 (0.74) | 2.47 (0.79) | -0.80 (0.86) | 2.11 (0.69) | 2.64 (0.86) | 1.38 (0.59) | -3.10 (0.83)

10. Secondary Outcome: Parts 1 and 2: Percent Change From Baseline in Triglycerides, High Density Lipoprotein (HDL) Cholesterol (c), Non-HDLc, LDLc, Hemoglobin (HbA1C), Alanine Transaminase, Aspartate Aminotransferase, N-terminal Propeptide of Type III Collagen (Pro-C3)
Description: LS Mean was calculated using MMRM.
Time Frame: Part 1: Baseline, Day 92; Part 2: Baseline, Day 141
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 6 | 12 | 11 | 10 | 14 | 9 | 19 | 20
Percent change
  Triglycerides: number analyzed (Participants) | 5 | 11 | 10 | 7 | 9 | 7 | 17 | 18
  Triglycerides | -22.74 (11.53) | -23.95 (7.74) | -17.71 (8.20) | -27.63 (9.66) | -28.49 (8.62) | -20.71 (9.74) | -2.21 (6.23) | -25.30 (5.66)
  HDLc: number analyzed (Participants) | 5 | 11 | 10 | 7 | 10 | 7 | 17 | 18
  HDLc | 18.17 (5.43) | 11.19 (3.68) | 9.20 (3.92) | 2.90 (4.50) | 20.10 (3.73) | 9.79 (4.56) | 1.96 (2.97) | 22.65 (5.58)
  Non HDLc: number analyzed (Participants) | 5 | 11 | 10 | 7 | 10 | 7 | 17 | 18
  Non HDLc | -6.31 (6.45) | -13.87 (4.61) | -1.92 (4.74) | -16.32 (5.51) | -7.75 (4.38) | -6.34 (5.39) | 1.18 (3.56) | -17.12 (3.53)
  LDLc: number analyzed (Participants) | 5 | 11 | 10 | 7 | 10 | 7 | 17 | 18
  LDLc | -6.17 (7.38) | -13.45 (5.29) | 2.59 (5.41) | -16.46 (6.34) | -5.02 (5.06) | -4.11 (6.20) | 1.15 (4.08) | -12.36 (4.80)
  HbA1C: number analyzed (Participants) | 5 | 11 | 10 | 7 | 13 | 7 | 18 | 19
  HbA1C | 7.36 (4.05) | 1.80 (2.84) | 3.05 (2.99) | -3.66 (3.42) | -1.85 (2.60) | 6.89 (3.43) | 0.61 (2.28) | -7.23 (1.66)
  Alanine Transaminase: number analyzed (Participants) | 4 | 11 | 10 | 7 | 13 | 7 | 18 | 19
  Alanine Transaminase | -16.87 (10.62) | -26.65 (6.99) | -26.73 (7.40) | -43.69 (8.55) | -18.83 (6.38) | -39.84 (8.42) | -4.18 (5.47) | -45.80 (3.86)
  Aspartate Aminotransferase: number analyzed (Participants) | 4 | 11 | 10 | 7 | 13 | 7 | 18 | 19
  Aspartate Aminotransferase | -29.36 (9.47) | -19.90 (6.15) | -15.10 (6.52) | -37.88 (7.52) | -11.41 (5.63) | -25.32 (7.43) | -4.40 (4.85) | -47.28 (3.54)
  Pro-C3: number analyzed (Participants) | 4 | 11 | 10 | 10 | 13 | 7 | 18 | 19
  Pro-C3 | -19.71 (14.53) | -18.79 (9.02) | 1.08 (9.38) | -27.67 (11.20) | -11.18 (8.19) | -12.76 (11.22) | 3.26 (7.02) | -19.52 (3.28)

11. Secondary Outcome: Part 1: Percent Change From Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) at Day 92
Description: LS Mean was calculated using MMRM. HOMA-IR value was calculated by multiplying fasting Glucose (mg/dL) with fasting Insulin (uIU/ml) and then dividing by 405.
Time Frame: Baseline, Day 92
Population: The analysis set included all randomized participants who received at least 1 dose of investigational product and who had measurable post-baseline PD data in Part 1. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W
Number analyzed (Participants) | 1 | 3 | 6 | 7 | 11 | 5 | 11
Percent change | 10.37 (51.30) | 7.40 (30.62) | 37.07 (20.87) | -41.42 (19.48) | -4.57 (15.57) | -41.11 (23.39) | -0.09 (15.72)

12. Secondary Outcome: Part 1: Percent Change From Baseline in Adiponectin at Day 92
Description: LS Mean was calculated using MMRM.
Time Frame: Baseline, Day 92
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W
Number analyzed (Participants) | 5 | 11 | 10 | 7 | 13 | 7 | 18
Percent change | 37.65 (14.48) | 25.46 (9.88) | 29.09 (10.47) | 60.85 (12.00) | 23.11 (9.07) | 24.14 (12.10) | -4.25 (7.80)

13. Secondary Outcome: Part 1: Percent Change From Baseline in Free Fatty Acid at Day 92
Description: LS Mean was calculated using MMRM.
Time Frame: Baseline, Day 92
Population: The analysis set included all randomized participants who received at least 1 dose of study intervention and who had measurable post-baseline PD data in Part 1. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W
Number analyzed (Participants) | 5 | 7 | 10 | 6 | 9 | 7 | 16
Percent change | 28.70 (24.68) | 50.20 (21.05) | 27.08 (17.76) | 51.58 (22.08) | 43.85 (18.17) | 56.12 (20.81) | 20.91 (13.96)

14. Secondary Outcome: Part 1: Percent Change From Baseline in Adipose Tissue Insulin Resistance (Adipo-IR) at Day 50
Description: LS Mean was calculated using MMRM. Adipo-IR was derived from fasting insulin and free fatty acid.
Time Frame: Baseline, Day 50
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 7 | 8 | 6 | 14
Percent change | -6.12 (61.71) | 82.00 (59.79) | 3.28 (60.01) | 78.40 (46.41) | -25.96 (42.75) | -10.36 (50.33) | -15.82 (32.62)

15. Secondary Outcome: Parts 1 and 2: Percent Change From Baseline in Liver Fat as Assessed Via Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF)
Description: LS Mean was calculated using MMRM.
Time Frame: Part 1: Baseline, Day 92; Part 2: Baseline, Day 141
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 5 | 11 | 10 | 7 | 13 | 8 | 18 | 19
Percent change | -36.94 (11.01) | -49.62 (7.73) | -36.11 (8.14) | -60.39 (9.40) | -43.19 (6.99) | -50.39 (9.07) | 9.77 (6.04) | -64.69 (3.38)

16. Secondary Outcome: Part 2: Number of Participants With at Least an Improvement of Fibrosis ≥1 Stage Without Worsening of NASH
Description: Fibrosis improvement was defined as ≥1-stage decrease in NASH CRN fibrosis score.
  Worsening of NASH was defined as increase ≥1 point in NAS for ballooning or inflammation.
  NASH CRN Fibrosis was staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: Day 141
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 19
Participants | 5

17. Secondary Outcome: Part 2: Number of Participants With NASH Resolution Without Worsening of Fibrosis
Description: Resolution of NASH included the total absence of ballooning (score=0) and absent or mild inflammation (score 0 to 1).
  Worsening of fibrosis was defined as progression of fibrosis ≥1 stage in NASH CRN fibrosis score.
  NASH CRN Fibrosis was staged on a 0-4 scale: 0 (none); 1 (perisinusoidal or periportal fibrosis); 2 (perisinusoidal and portal/periportal fibrosis); 3 (bridging fibrosis); 4 (cirrhosis).
Time Frame: Day 141
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Pegozafermin 27 mg QW
Number analyzed (Participants) | 19
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were collected after dosing to end of study (up to 113 days for Part 1 and up to 162 days for Part 2).
Description: The Safety Analysis set included all randomized participants who received at least 1 dose of study intervention. Arm groups were based upon the actual treatment received for the purpose of safety analysis.
  MedDRA version 23.0 was used for Part 1 and MedDRA version 23.1 was used for Part 2.
Arm/Group | Part 1: Pegozafermin 3 mg QW | Part 1: Pegozafermin 9 mg QW | Part 1: Pegozafermin 18 mg QW | Part 1: Pegozafermin 27 mg QW | Part 1: Pegozafermin 18 mg Q2W | Part 1: Pegozafermin 36 mg Q2W | Part 1: Placebo QW or Q2W | Part 2: Pegozafermin 27 mg QW
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12 | 0/11 | 0/10 | 0/14 | 0/9 | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12 | 0/11 | 0/10 | 1/14 | 1/9 | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 6/7 | 4/12 | 7/11 | 7/10 | 8/14 | 8/9 | 8/18 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pegozafermin 3 mg QW (N=7) | Part 1: Pegozafermin 9 mg QW (N=12) | Part 1: Pegozafermin 18 mg QW (N=11) | Part 1: Pegozafermin 27 mg QW (N=10) | Part 1: Pegozafermin 18 mg Q2W (N=14) | Part 1: Pegozafermin 36 mg Q2W (N=9) | Part 1: Placebo QW or Q2W (N=18) | Part 2: Pegozafermin 27 mg QW (N=20)
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pegozafermin 3 mg QW (N=7) | Part 1: Pegozafermin 9 mg QW (N=12) | Part 1: Pegozafermin 18 mg QW (N=11) | Part 1: Pegozafermin 27 mg QW (N=10) | Part 1: Pegozafermin 18 mg Q2W (N=14) | Part 1: Pegozafermin 36 mg Q2W (N=9) | Part 1: Placebo QW or Q2W (N=18) | Part 2: Pegozafermin 27 mg QW (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bundle Branch Block Left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid Mass (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Change of Bowel Habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 1 | 2 | 4 | 7
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 10
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 4
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Injection Site Bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injection Site Erythema (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Injection Site Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Swelling Face (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Enzyme Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 4 | 2 | 0 | 2 | 2 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT04048135/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04048135/SAP_001.pdf